CLINICAL TRIAL: NCT04176900
Title: 3D Printed Rigid Bolus Versus Silicone Bolus: A Comparative Study
Brief Title: 3D Printed Rigid Bolus Versus Silicone Bolus for Treatment of Tumors Involving the Skin: A Comparative Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed during Covid Pandemic, and no longer supported locally
Sponsor: Nova Scotia Cancer Centre (Other)
Responsible Party: Principal Investigator, Lara Best, MD, FRCPC, MMEd, Radiation Oncologist, Nova Scotia Cancer Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15441
Record Dates: First submitted 2019-11-22; First posted 2019-11-25 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Skin Neoplasm Malignant; Skin Cancer
Keywords: Radiation Therapy; Radiation Dosimetry; Patient Reported Outcomes; 3D-printed bolus
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will have both the rigid and flexible 3D printed boluses made. Each will be used on alternate days during radiation therapy treatments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alternating 3D boluses (Experimental): Both rigid and flexible 3D printed boluses made for each patient. Each is used on alternate days during radiation therapy.
  Interventions: Other: Ingeo Biopolymer (PLA); Other: Ecoflex 030

INTERVENTIONS:
Other: Ingeo Biopolymer (PLA) — Biopolymer used for 3D-printing of rigid bolus
  Other Names: 3D-Fuel PLA
Other: Ecoflex 030 — Polymer used for the 3D-printed flexible bolus
  Other Names: Body Double & Body Double SILK; Dragon Skin Series & F/X Pro; Encapso K; Equinox Series; EZ Brush Silicone; EZ-Spray Silicone Series; Mold Max Series; Mold Star Series; OOMOO Series; PoYo Putty 40; Psycho Paint; Rebound Series; Rubber Glass; Silicone 1515, 1603, 3030, 1708; Skin Tite; Smooth-Sil Series; Solaris; SomaFoama Series; SORTA-Clear Series

SUMMARY:
This study compares two types of 3D-printed skin bolus (rigid and flexible) used to optimize the treatment of tumors/cancers involving the skin. Each patient will have both types of bolus made, with each will be used on alternating days. The goal is to determine if one type of bolus provides a better fit and thus radiotherapy plan, the ease of use of each type of bolus, and patient reported feedback.

DETAILED DESCRIPTION:
Need for Skin Bolus during Radiotherapy for Cancers that Involve the Skin Using standard megavoltage (MV) radiotherapy to treat tumors that involve the skin is technically challenging as without modification, the high-energy radiotherapy machines under-dose the superficial tissue. This is a problem, as this may lead to an inadequate radiation dose being delivered to the skin, thus compromising tumor control. To compensate for this, a flexible polymer material ("bolus") measuring 5-10mm in thickness is placed over the skin during radiotherapy.

There are many types of boluses used internationally from rubber to candle wax slabs. The bolus allows the radiation dose to build up so that a sufficient dose is deposited at the skin. Use of bolus for cancers involving the skin is considered the standard of care when using conventional MV radiotherapy.

Challenges of Using Conventional Bolus Many standard boluses are slightly flexible, but are not able to follow significant changes in the underlying contours. When a bolus is not able to follow an individual's unique 'peaks and valleys' in contour, it can lead to air gaps between the bolus and the skin. An air gap, which is easily seen during imaging, can also vary on a day-to-day basis due to slight changes in positioning of the bolus prior to radiotherapy treatment. The varying air gaps can affect how much radiation dose is getting to the skin, and can potentially lead to under-dosing of the cancer cells in the skin. Even small air gaps (i.e. 5mm in thickness), can cause a 5% error in dose, which exceeds the safe tolerance for treatment.

Areas where this can be a problem are where the patient's anatomy undergoes significant topographical changes in a small area. Examples of this include the ear, nose, top of head. Patients with metastatic cancer can also have large lymph nodes or masses that are growing towards the skin that can be difficult to accommodate with standard bolus materials.

3D-Printed Bolus One method to overcome challenging anatomy for cases that require skin bolus for radiotherapy is the use of 3D-printed bolus. This technology uses data acquired from a CT scan of the affected area. The patients contour can then be used to create an individualized bolus that matches the patient contour for the treatment field. This technology has been demonstrated to improve fit (less air gaps) and decreased radiotherapy treatment time. The bolus used in this study was rigid.

Trial design and Rationale Other than the chestwall study, the literature on 3D-printed bolus for radiotherapy has focused on the dosimetry and feasibility of using this technology. However, it is used in an ad hoc method in many centers, using various workflows. There are no studies examining which type of bolus provides the best radiotherapy plan, is the easiest to use at the radiation therapy machines or which is preferred by patients.

To fill this gap, this study will aim to answer a few questions. It will compare the use of rigid 3D-printed bolus (most commonly used and reported in the literature) versus a flexible silicone 3D-printed bolus. Both types of bolus will be used to treat patients with cancers involving the skin. This will allow comparison of radiotherapy plans for each patient between the two types of bolus where each subject is his/her own control. The study will also collect data about real-time set-up using each bolus and feedback from radiation therapists (deliver radiation treatments) about the ease of use of each. Lastly, patients will complete a short survey to provide feedback about comfort with use of each type of bolus and to determine if one type of bolus is favored over the other.

This data will be instrumental is determining the standard of care of the use of 3D-printed bolus as it will assess two types of bolus in three domains: ability to help generate an adequate radiotherapy plan, ease of use by the specialists that deliver the radiotherapy (radiation therapists) and patient reported feedback.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of a primary skin cancer or metastatic cancer with involvement of the skin or underlying soft tissues
* Being treated with radiation therapy that requires the use of bolus to ensure adequate radiotherapy dose to the skin in the affected area
* Planned for palliative or curative intent radiotherapy using megavoltage (MV) photons
* Site of involvement has significant contour change, leading to anticipated challenges using conventional bolus material
* Patient must be competent and able to complete informed consent
* Age ≥ 18
* Women of childbearing potential must be proven to not be pregnant or breast feeding

Exclusion Criteria:

* Patient being treated with a radiotherapy technique that does not require bolus
* Patient being treated with a radiotherapy technique other than MV photons (i.e. electrons, brachytherapy, kilovoltage (kV) photons)
* Patient of childbearing potential who is pregnant, actively trying to become pregnant or breast feeding
* Allergy to silicone or other components of either the 3D printed rigid or flexible bolus.
* Size of the bolus required for treatment exceeds 25cm in maximum diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Air Gap measurement | 6 weeks
  Measurement of the gap between the bolus and the surface of the patient
Planned versus expected radiation duse | 6 weeks
  Comparison of the planned radiation dose at skin, and that measured during radiation therapy treatment

SECONDARY OUTCOMES:
Ease of Use | 6 weeks
  Time required to place bolus in proper location prior to each radiation therapy treatment
Radiation Therapist ease of use | 6 weeks
  Radiation therapists asked to rate ease of use for each type of bolus
Challenges with Bolus Use | 6 weeks
  Comparison of the number of times each bolus could not be adequately applied prior to radiation therapy treatment
Patient Reported Outcomes | 6 weeks
  Patients asked about comfort associated with each bolus, their preference between the two, and any other feedback on the boluses
Fabrication time | 2 weeks
  Comparison of average fabrication time for each type of bolus
Successful fabrication | 2 weeks
  Comparison of percentage of cases for which an acceptable bolus could be created for each type of bolus

CONTACTS AND LOCATIONS:
Overall Officials: Lara R Best, MD, FRCPC, Principal Investigator — Nova Scotia Cancer Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canters RA, Lips IM, Wendling M, Kusters M, van Zeeland M, Gerritsen RM, Poortmans P, Verhoef CG. Clinical implementation of 3D printing in the construction of patient specific bolus for electron beam radiotherapy for non-melanoma skin cancer. Radiother Oncol. 2016 Oct;121(1):148-153. doi: 10.1016/j.radonc.2016.07.011. Epub 2016 Jul 27. PMID 27475278
- [Background] Dipasquale G, Poirier A, Sprunger Y, Uiterwijk JWE, Miralbell R. Improving 3D-printing of megavoltage X-rays radiotherapy bolus with surface-scanner. Radiat Oncol. 2018 Oct 19;13(1):203. doi: 10.1186/s13014-018-1148-1. PMID 30340612
- [Background] Kong Y, Yan T, Sun Y, Qian J, Zhou G, Cai S, Tian Y. A dosimetric study on the use of 3D-printed customized boluses in photon therapy: A hydrogel and silica gel study. J Appl Clin Med Phys. 2019 Jan;20(1):348-355. doi: 10.1002/acm2.12489. Epub 2018 Nov 7. PMID 30402935
- [Background] Robar JL, Moran K, Allan J, Clancey J, Joseph T, Chytyk-Praznik K, MacDonald RL, Lincoln J, Sadeghi P, Rutledge R. Intrapatient study comparing 3D printed bolus versus standard vinyl gel sheet bolus for postmastectomy chest wall radiation therapy. Pract Radiat Oncol. 2018 Jul-Aug;8(4):221-229. doi: 10.1016/j.prro.2017.12.008. Epub 2017 Dec 24. PMID 29452866
- See also: National Comprehensive Cancer Network (NCCN). Squamous Cell Skin Cancer. NCCN Clinical Practice Guidelines in Oncology. Version 1.2020. — https://www.nccn.org/professionals/physician_gls/pdf/squamous.pdf